CLINICAL TRIAL: NCT05623098
Title: Effects of Dietary Fiber Enteral Nutrition on Bone Metabolism in Septic Patients
Brief Title: Effects of Dietary Fiber on Bone Metabolism
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Cuiping Liu, Chief researcher, Zhujiang Hospital
Other Study IDs: 2022LX0036_GC
Record Dates: First submitted 2022-08-31; First posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Sepsis
Keywords: short-chain fatty acid; sepsis; bone metabolism
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dietary fiber was not added to enteral nutrition preparation: Dietary fiber was not added to enteral nutrition preparation
- Dietary fiber was added to enteral nutrition preparation: Dietary fiber was added to enteral nutrition preparation
  Interventions: Dietary Supplement: dietary fiber nutrients

INTERVENTIONS:
Dietary Supplement: dietary fiber nutrients — Whether to add nutrients containing dietary fiber
  Groups: Dietary fiber was added to enteral nutrition preparation

SUMMARY:
Clinical and animal studies have found that sepsis can lead to a serious imbalance in the gut microecology, a reduction in probiotics, a reduction in short-chain fatty acid, a reduction in bone mass, and an increase in bone destruction, maintaining the stability of microecology can be one of the effective means of bone protection. But at present, the treatment of sepsis with early supplementation of probiotics is still controversial, and dietary fiber intake has significantly changed the composition of the microbiota, it may be a safe and effective method to prevent bone loss in sepsis. Further study on it will provide reliable theoretical basis and intervention target for early, safe and effective prevention of osteoporosis.

DETAILED DESCRIPTION:
In recent years, researchers have found that the incidence of bone loss in ICU patients is significantly higher than that in the control group of the same age, patients with sepsis whose bone balance is disrupted by higher overresorption, bone destruction and release of multiple active cytokines and toxins become the"Invisible killer"of the ICU, however, the pathogenesis of osteoporosis is not clear, and the existing drugs for osteoporosis can not be safely used in critically ill patients. The gastrointestinal tract is the"Initiating organ"and"Central organ" of multiple organ dysfunction and forms a complex and powerful"Gut-bone axis"with bone, which plays a key role in bone metabolism, but the mechanism is unclear. The human gut contains a dense and diverse microbial community, which plays an important role in nutrition, metabolism and immunity, small intestinal microecology can affect bone turnover through a variety of pathways, especially the metabolite short-chain fatty acid FAS (SCFAs) , which can inhibit osteoclast activity by regulating inflammatory cytokines and immune cells, promote the formation of osteoblasts and other aspects to maintain the stability of bone metabolism, and then protect the health of bones, forming a"Gut-microcology-bone"axis.

Clinical and animal studies have found that sepsis can lead to a serious imbalance in the gut microecology, a reduction in probiotics, a reduction in short-chain fatty acid, a reduction in bone mass, and an increase in bone destruction, maintaining the stability of microecology can be one of the effective means of bone protection. But at present, the treatment of sepsis with early supplementation of probiotics is still controversial, and dietary fiber intake has significantly changed the composition of the microbiota, it may be a safe and effective method to prevent bone loss in sepsis. Further study on it will provide reliable theoretical basis and intervention target for early, safe and effective prevention of osteoporosis. Therefore, based on the above research background, Investigators intend to evaluate the overall safety and efficacy of dietary fiber-containing enteral nutrition supplementation in patients with sepsis by observing changes in bone metabolism-related indicators, to provide the basis for further basic and mechanism research

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily cooperated with the study and signed the informed consent form, and could be followed up
2. Age 18-70
3. It meets the diagnostic criteria of Sepsis 2016 Sepsis 3.0 guidelines
4. After treatment, the Hemodynamics is stable and the patient is ready to start enteral nutrition support
5. Those who need tube feeding for more than 14 days because of the need of illness and can not take food by mouth

Exclusion Criteria:

1. People who have had osteoporosis in the past
2. Admission due to fracture
3. The shock was not corrected, and the patients were maintained with a large amount of vaso-active drugs (0.5 ug/kg/min of noradrenaline) , but could not be given enteral nutrition
4. Supplement with probiotics or prebiotics alone
5. Parturients
6. No written informed consent

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1) sepsis 20163.0: infection + sequential organ failure assessment (Sofa) score ≥2 points. (rapid SOFA (qSOFA) scoring tool criteria: (1) respiratory frequency ≥22 beats/min; (2) change in state of consciousness; (3) systolic blood pressure ≤100 mm Hg) .
Sampling Method: Non-Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The changes of bone metabolic markers β-CTX | 28 day
  The venous blood was drawn daily before and after the enrollment (the first, third, seventh and fourteenth days) ，and β- CTX for comparison
The changes of bone metabolic markers PINP | 28 day

SECONDARY OUTCOMES:
Changes in intestinal flora | 28 day
  Collect stool before and after the enrollment (the first, third, seventh and fourteenth days) ，observe the changes of intestinal flora in the two groups. Total bacterial DNA were extracted from samples using the QIAamp DNA stool Mini Kit from Qiagen according to the manufacture's protocol.
Changes in short-chain fatty acid of metabolites | 28 day
  Collect stool before and after the enrollment (the first, third, seventh and fourteenth days) ，observe the changes of metabolite short chain fatty acids in the two groups. Fresh feces were collected and frozen in liquid nitrogen timely.SCFAs was extracted and quantified using a Metrohm ion chromatograph(850 Professional Ic, Metrohm, Herisau, Switzerlan) system
Abdominal symptoms (abdominal distention) | 28 day
  To evaluate and compare the difference of abdominal symptoms (abdominal distension) between the two groups，It is divided into three levels according to the severity of abdominal distension, it can be divided into light, medium and severe (for example:Mild, soft abdomen, tolerable，Moderate: abdominal bulge, obvious discomfort，Severe: abdominal muscles are obviously tense/intolerable)
Abdominal symptoms ( diarrhea incidence) | 28 day
  To evaluate and compare the difference of abdominal symptoms (diarrhea incidence ) between the two groups，it can be divided into light, medium and severe (for example:Mild, 3-5 times/day, 250-500ml/day，Moderate:>5 times/day, 500-1000ml/day,Severity:>5 times/day,>1500ml/day)
The change of systemic inflammatory response index: the value of TNF-α in systemic inflammatory response | 28 day
  The changes of TNF-α were observed and compare before and after treatment, It can be tested in the laboratory of our hospital, the higher the value, the heavier the infection.
The change of systemic inflammatory response index: the value of IL-6 in systemic inflammatory response | 28 day
  The changes of IL-6 were observed and compare before and after treatment. It can be tested in the laboratory of our hospital, the higher the value, the heavier the infection
The change of systemic inflammatory response index: the value of Procalcitonin in systemic inflammatory response | 28 day
  The changes of procalcitonin were observed and compare before and after treatment, the higher the value, the heavier the infection
Length of ICU stay | 28 day
  The total hospitalization time were observed before and after treatment
Length of Apache II score | 28 day
  The total Apache II score were observed before and after treatment，The higher the score is, the more serious the disease is.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang hospital, Guangzhou, Guangdong, China